CLINICAL TRIAL: NCT02181504
Title: A Study of Abicipar Pegol in Japanese Patients With Neovascular Age-related Macular Degeneration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 150998-002; BAMBOO (Other: Allergan)
Record Dates: First submitted 2014-07-02; First posted 2014-07-04 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-03

CONDITIONS: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — abicipar pegol; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- abicipar pegol 2 mg (Experimental): Abicipar pegol 2 mg administered to the study eye by intravitreal injection at day 1, weeks 4 and 8, followed by a sham procedure at weeks 12 and 16.
  Interventions: Drug: abicipar pegol; Other: sham procedure
- abicipar pegol 1 mg (Experimental): Abicipar pegol 1 mg administered to the study eye by intravitreal injection at day 1, weeks 4 and 8, followed by a sham procedure at weeks 12 and 16.
  Interventions: Drug: abicipar pegol; Other: sham procedure
- ranibizumab 0.5 mg (Active Comparator): Ranibizumab (Lucentis®) 0.5 mg administered to the study eye by intravitreal injection every 4 weeks from day 1 through week 16.
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: abicipar pegol — Abicipar pegol administered to the study eye by intravitreal injection at day 1, weeks 4 and 8.
  Arms: abicipar pegol 1 mg; abicipar pegol 2 mg
Drug: ranibizumab — Ranibizumab (Lucentis®) 0.5 mg administered to the study eye by intravitreal injection every 4 weeks from day 1 through week 16.
  Other Names: Lucentis®
  Arms: ranibizumab 0.5 mg
Other: sham procedure — Sham procedure to the study eye at weeks 12 and 16.
  Arms: abicipar pegol 1 mg; abicipar pegol 2 mg

SUMMARY:
This is a safety and efficacy study of abicipar pegol in patients with neovascular age-related macular degeneration to establish comparability between Japanese and non-Japanese.

ELIGIBILITY:
Inclusion Criteria:

* Ethnically Japanese
* Diagnosis of wet age-related macular degeneration in at least 1 eye
* Best corrected visual acuity of 20/32 to 20/320 in the study eye and 20/200 or better in the fellow eye

Exclusion Criteria:

* Hypersensitivity, allergy, or anaphylactic reaction to iodine or shellfish
* Cataract or refractive surgery within the last 3 months
* History of vitrectomy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (11):
- Japan (11):
  - Nihon University Hospital, Chiyoda-ku,Tokyo
  - 1 Fukushima Medical University, Fukushima
  - Kyushu University Hospital, Kita-ku, Fukuoka-shi Fukuoka
  - Okayama University Hospital, Kita-ku, Okayama-shi Okayama
  - Shiga University, Ōtsu
  - Tokyo Women's Medical University, Shinjuku-ku
  - Nagoya University Hospital, Showa-ku, Nagoya-shi Aichi
  - Takeuchi Eye Clinic, Taito Ku Tokyo
  - Musashi Dream Clinic, Tennoji-ku Osaka
  - Juntendo University Urayas, Urayasu-shi
  - Otakeganka Tsukimino Clinic, Yamato Kanagawa

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Abicipar Pegol 2 mg | Abicipar Pegol 1 mg | Ranibizumab 0.5 mg
Started | 10 | 10 | 5
Completed | 9 | 9 | 4
Not Completed | 1 | 1 | 1
Not completed — Adverse Event | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abicipar Pegol 2 mg | Abicipar Pegol 1 mg | Ranibizumab 0.5 mg | Total
Number analyzed (Participants) | 10 | 10 | 5 | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.8 (5.75) | 75.6 (7.18) | 76.6 (9.24) | 74.3 (7.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 4
  Male | 8 | 9 | 4 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) in the Study Eye
Description: BCVA is measured using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase (positive number change from baseline) in the number of letters read correctly means that vision has improved and a decrease (negative number change from baseline) in the number of letters read correctly means that vision has worsened.
Time Frame: Baseline, Week 16
Population: Modified Intent-to-Treat: all randomized and treated patients with at least 1 follow-up visit
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Abicipar Pegol 2 mg | Abicipar Pegol 1 mg | Ranibizumab 0.5 mg
Number analyzed (Participants) | 10 | 10 | 5
Letters
  Baseline | 58.5 (17.30) | 54.3 (15.58) | 55.8 (9.68)
  Change from Baseline at Week 16 | 8.9 (9.16) | 7.8 (8.51) | 17.4 (8.08)

2. Secondary Outcome: Change From Baseline in BCVA in the Study Eye
Description: as for outcome 1
Time Frame: Baseline, Week 20
Population: Modified Intent-to-Treat: all randomized and treated patients with at least 1 follow-up visit
Measure: Mean (Standard Deviation); unit: Letters
Groups:
- Abicipar Pegol 2 mg; Abicipar Pegol 1 mg: Abicipar pegol 1 mg administered to the study eye by intravitreal injection at day 1, weeks 4 and 8, followed by a sham procedure at weeks 12 and 16.
Arm/Group | Abicipar Pegol 2 mg | Abicipar Pegol 1 mg | Ranibizumab 0.5 mg
Number analyzed (Participants) | 10 | 10 | 5
Letters
  Baseline | 58.5 (17.30) | 54.3 (15.58) | 55.8 (9.68)
  Change from Baseline at Week 20 | 9.6 (6.75) | 8.7 (7.33) | 17.2 (7.73)

3. Secondary Outcome: Percentage of Patients With a BCVA Gain of ≥15 Letters in the Study Eye on the Early Treatment Diabetic Retinopathy Study (ETDRS) Scale
Description: BCVA is measured using an eye chart and is reported as the number of letters read correctly using the ETDRS Scale (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved. The percentage of patients with a BCVA gain of ≥15 letters are noted.
Time Frame: Baseline, 20 Weeks
Population: Modified Intent-to-Treat: all randomized and treated patients with at least 1 follow-up visit
Measure: Number; unit: Percentage of Patients
Arm/Group | Abicipar Pegol 2 mg | Abicipar Pegol 1 mg | Ranibizumab 0.5 mg
Number analyzed (Participants) | 10 | 10 | 5
Percentage of Patients | 20.0 | 30.0 | 60.0

4. Secondary Outcome: Percentage of Patients With a BCVA Gain of ≥10 Letters in the Study Eye on the ETDRS Scale
Description: BCVA is measured using an eye chart and is reported as the number of letters read correctly using the ETDRS Scale (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved. The percentage of patients with a BCVA gain of ≥10 letters are noted.
Time Frame: Baseline, 20 Weeks
Population: Modified Intent-to-Treat: all randomized and treated patients with at least 1 follow-up visit
Measure: Number; unit: Percentage of Patients
Arm/Group | Abicipar Pegol 2 mg | Abicipar Pegol 1 mg | Ranibizumab 0.5 mg
Number analyzed (Participants) | 10 | 10 | 5
Percentage of Patients | 50.0 | 50.0 | 80.0

5. Secondary Outcome: Change From Baseline in Central Retinal Thickness (CRT) in the Study Eye
Description: CRT is assessed using spectral domain optical coherence tomography (SD-OCT), a non-invasive diagnostic system that provides high-resolution imaging sections of the retina. SD-OCT is performed in the study eye after pupil dilation. A negative change from Baseline indicates improvement and a positive change from baseline indicates worsening.
Time Frame: Baseline, Week 16, Week 20
Population: Modified Intent-to-Treat: all randomized and treated patients with at least 1 follow-up visit
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Abicipar Pegol 2 mg | Abicipar Pegol 1 mg | Ranibizumab 0.5 mg
Number analyzed (Participants) | 10 | 10 | 5
microns
  Baseline | 438.7 (107.32) | 475.1 (192.76) | 470.0 (67.75)
  Change from Baseline at Week 16 | -196.5 (124.20) | -187.3 (145.63) | -230.4 (59.28)
  Change from Baseline at Week 20 | -194.9 (109.37) | -139.4 (110.66) | -250.6 (50.69)

ADVERSE EVENTS:
Description: The Safety Population included all enrolled patients and is used to assess adverse events and serious adverse events.
Arm/Group | Abicipar Pegol 2 mg | Abicipar Pegol 1 mg | Ranibizumab 0.5 mg
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 2/5
Other Adverse Events (participants affected / at risk) | 4/10 | 8/10 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abicipar Pegol 2 mg (N=10) | Abicipar Pegol 1 mg (N=10) | Ranibizumab 0.5 mg (N=5)
Cataract (Eye disorders) | 0 | 0 | 1
Angle closure glaucoma (Eye disorders) | 0 | 0 | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Embolic stroke (Nervous system disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abicipar Pegol 2 mg (N=10) | Abicipar Pegol 1 mg (N=10) | Ranibizumab 0.5 mg (N=5)
Iritis (Eye disorders) | 1 | 1 | 0
Vitreous floaters (Eye disorders) | 1 | 1 | 0
Vitreous opacities (Eye disorders) | 1 | 1 | 0
Foreign body sensation in eyes (Eye disorders) | 1 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 4 | 0
Cataract (Eye disorders) | 0 | 1 | 0
Anterior chamber inflammation (Eye disorders) | 0 | 1 | 0
Asthenopia (Eye disorders) | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0
Device breakage (General disorders) | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 1 | 0
Eosinophil count increased (Investigations) | 0 | 1 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Injection site haemorrhage (General disorders) | 0 | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Periodontitis (Infections and infestations) | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0
Vitritis (Eye disorders) | 0 | 1 | 0
Intraocular pressure increased (Investigations) | 0 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Retinal exudates (Eye disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If the site intends to publish the Clinical Trial results and other information with an academic intention, or Allergan intends to utilize the related information for distribution activities of its own, the said party must obtain the consent from the other party in advance. However, except for the case based on the due reason including that the consent of trial subjects cannot be obtained though it is mandatory, the other party cannot refuse the consent.